CLINICAL TRIAL: NCT05843578
Title: A Phase 2a, Randomized, Placebo-controlled, Double-blind Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of AGMB-129 in Patients With Fibrostenotic Crohn's Disease
Brief Title: STENOVA - A Study to Evaluate Safety, Tolerability, PK and PD of AGMB-129 in Patients With Fibrostenotic Crohn's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Agomab Spain S.L.U. (Industry)
Responsible Party: Sponsor
Organization: Agomab Therapeutics NV (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGMB-129-C102
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Fibrostenotic Crohn's Disease

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, parallel, multicenter, phase 2a study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AGMB-129 High (Experimental): AGMB-129 high dose
  Interventions: Drug: AGMB-129
- AGMB-129 Low (Experimental): AGMB-129 low dose
  Interventions: Drug: AGMB-129
- Placebo (Experimental): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AGMB-129 — Oral capsule
  Arms: AGMB-129 High; AGMB-129 Low
Drug: Placebo — Matching oral capsule
  Arms: Placebo

SUMMARY:
Many patients with Crohn's disease develop fibrotic narrowing (strictures) in their bowel, causing obstructive symptoms such as abdominal pain, cramping, or vomiting after meals. Because of these symptoms, patients often require bowel resection surgery. The objective of this clinical trial is to evaluate the safety, pharmacokinetics, and pharmacodynamics of AGMB-129 in patients with Crohn's disease and symptomatic strictures, and whether it can have a beneficial effect on intestinal strictures.

The participants will be in the Part A for a duration of up to 19 weeks including a 5 week screening period, a 12-week double-blind, placebo-controlled treatment period, and 2 week safety follow up period. Participants who continue to Part B can receive treatment for up to an additional 48 weeks, with a safety follow-up visit 2 weeks after the last dose of treatment.

DETAILED DESCRIPTION:
Part A is a randomized, placebo-controlled, double-blind, parallel, multicenter, phase 2a study in participants with Crohn's disease and symptomatic intestinal strictures.

Part A consists of 3 periods (a screening period, a placebo-controlled, double-blind treatment period, and safety follow-up). After signing informed consent, eligibility will be assessed during a 5-week screening period. The presence of qualifying intestinal strictures will be assessed by ileocolonoscopy and magnetic resonance enterography (MRE). The presence of obstructive symptoms will be also evaluated.

Eligible participants will be randomized 1:1:1 to receive AGMB-129 high dose, low dose or placebo for 12 weeks.

During Screening and Week 12 visits, participants will undergo ileocolonoscopy with biopsy collection for exploring pharmacodynamics. Participants will have blood sample collection at Weeks 2, 4, 8, and 12 to assess safety, pharmacokinetics, and pharmacodynamics.

Throughout the study, participants will undergo routine safety assessments at study visits, which will include physical examination, vital signs, clinical laboratory assessment, electrocardiogram (ECG), and recording of AEs.

Part B is an open-label treatment extension for participants who have completed the double-blind treatment period in Part A.

ELIGIBILITY:
Inclusion Criteria (Part A):

1. Diagnosis of ileal or ileocolonic CD based on supporting guideline criteria (eg, clinical, endoscopic, and histologic evidence) established at least 3 months prior to screening.
2. Presence of at least 1 stricture in the terminal ileum within reach of an endoscope (passable or nonpassable).Strictures should be noncritical, naïve or anastomotic stricture(s), caused by CD and confirmed centrally by MRE according to the following criteria:

   * Localized luminal narrowing (luminal diameter ≤50% relative to normal adjacent bowel); AND
   * Bowel wall thickening (≥25% relative to adjacent bowel; AND
   * Either prestenotic dilation (defined as a luminal diameter ≥3 cm) or nonpassable with adult colonoscope
3. Presence of tolerable obstructive symptoms, as defined by a screening S-PRO severity score ≥2, and not expected to require hospitalization, endoscopic balloon dilation, surgical resection, or additional therapy during the study. Participant should have sufficient food intake, even with diet modification.
4. Stable background therapy for CD and agree to maintain background therapy for the study duration

Exclusion criteria (Part A):

1. History or current diagnosis of ulcerative colitis, indeterminate colitis, ischemic colitis, nonsteroidal anti-inflammatory drug-induced colitis, idiopathic colitis (ie, colitis not consistent with CD), radiation colitis, microscopic colitis, colonic mucosal dysplasia, or untreated bile acid malabsorption.
2. CD-related complications (previous extensive small bowel resection, ileorectal anastomosis, proctocolectomy, short bowel syndrome, ileostomy [diverting or end], colostomy, small bowel stoma, ileoanal pouch, inactive fistulae in or adjacent to an ileal stricture, anal and perianal stricture, active intra-abdominal or perianal abscess that has not been appropriately treated, abscess in relation to the stricture, toxic megacolon, very severe inflammation, or presence of deep ulceration in the colon or terminal ileum).
3. Ileitis not associated with CD (eg, ileitis associated with infections, spondyloarthropathies, ischemia, etc.).
4. Endoscopic balloon dilation or surgical treatment of the same small bowel stricture within the last 6 months prior to screening
5. Receiving cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil within 8 weeks of screening or Janus kinase inhibitor therapy within 4 weeks of screening.
6. Requiring continued treatment with systemically administered medications that are sensitive CYP3A4/5 substrates with a narrow therapeutic index or strong inhibitors of aldehyde oxidase or xanthine oxidase.
7. Current or history of vasculitis, valvulopathy or large vessel disorder or major abnormalities documented by cardiac echocardiography with Doppler

Inclusion Criteria (Part B):

1. Completion of the 12-week treatment period (Part A) and participant is willing and able to continue treatment.
2. Per investigator judgment, participant is able to continue or resume treatment following completion of the Week 12 visit in Part A.

Exclusion criteria (Part B):

1. More than 24 weeks since completion of the Week 12 visit in Part A.
2. Experienced any AE leading to permanent treatment discontinuation during treatment with study drug in the double blind treatment period (Part A).
3. Have undergone endoscopic balloon dilation or bowel surgery (resection surgery or strictureplasty) for any intestinal stricture since the Week 12 visit in Part A.
4. Developed any condition which meets the Part A exclusion criteria, as per investigator judgment.
5. Any condition which in the opinion of the investigator affects the safety or ability to participate in Part B.
6. Participation in any other clinical trial since the completion of the Week 12 visit in Part A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (Part A and B) | From Screening to Week 48
  To evaluate the safety and tolerability of AGMB-129 between AGMB-129 participants and placebo participants in terms of adverse events at every visit
Number of participants with abnormal clinical laboratory values (Part A and B) | From Screening to Week 48
  To evaluate the safety and tolerability of AGMB-129 between AGMB-129 participants and placebo participants in terms of abnormal laboratory parameters at every visit
Number of participants with abnormal ECG parameters (Part A and B) | From Screening to Week 48
  To evaluate the safety and tolerability of AGMB-129 between AGMB-129 participants and placebo participants in terms of abnormal ECG parameters at every visit
Number of participants with abnormal vital signs (Part A and B) | From Screening to Week 48
  To evaluate the safety and tolerability of AGMB-129 between AGMB-129 participants and placebo participants in terms of vital signs at every visit
Number of participants with abnormal physical exams (Part A and B) | From Screening to Week 48
  To evaluate the safety and tolerability of AGMB-129 between AGMB-129 participants and placebo participants in terms of physical exams at every visit
Number of participants with abnormal 2D-echocardiography (Part A and B) | From Screening to Week 48
  To evaluate the safety and tolerability of AGMB-129 between AGMB-129 participants and placebo participants in terms of echocardiography at week 12

SECONDARY OUTCOMES:
Plasma levels of AGMB-129 and its metabolites (Part A and B) | From Baseline to Week 48
  To characterize the pharmacokinetics (PK) of AGMB-129 and its metabolites by measuring the amount in plasma
Changes in mRNA gene expression in ileal biopsies ((Part A) | From Baseline to Week 48
  To characterize the pharmacodynamics of AGMB-129 by determining the gene expression in ileal biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Wiesel, MD, Study Director — Agomab Therapeutics
Locations (52):
- United States (11):
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - University of Miami, Miami, Florida
  - Digestive and Liver Center of Florida, Orlando, Florida
  - Gastroenterology Health Partners, New Albany, Indiana
  - Gastroenterology Health Partners, Louisville, Kentucky
  - Louisiana Research Center, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Gastro One, Cordova, Tennessee
- Austria (4):
  - Medical University of Graz, Graz
  - Gemeinnutzige Salzburger Landeskliniken Betriebsgesellschaft mbH (Landeskrankenhaus Salzburg/Regional Hospital Salzburg), Salzburg
  - Medical University Of Vienna (AKH Wien), Vienna
  - Hospital Landstrasse, Department of Internal Medicine IV, Vienna
- Canada (7):
  - University of Calgary, Calgary
  - Gastroenterology and Internal Medicine Research Institute (GIRI), Edmonton
  - South Edmonton Gastroenterology Research Clinic, Edmonton
  - Nova Scotia Health Authority, Halifax
  - TIDHI Innovation Inc., North York
  - Ottawa Hospital Research Institute, Ottawa
  - (G.I.R.I) GI Research Institute, Vancouver
- Denmark (5):
  - Aarhus University Hospital, Department of Hepatology and Gastroenterology, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Rigshospitalet - University Hospital Copenhagen, Copenhagen
  - Herlev Hospital (University of Copenhagen), Herlev
  - Odense University Hospital, Odense
- Germany (4):
  - Charite Universitatsmedizin Berlin KöR Campus Benjamin Franklin Medizinische, Berlin
  - Servicegesellschaft Krankenhaus Waldfriede mbH Krankenhaus Waldfriede e.V Akademisches Lehrkrankenhaus der Charite, Berlin
  - BSF Studiengesellschaft UG (Unternehmergesellschaft, haftungsbeschränkt), Halle
  - Universitatsklinikum Ulm AöR (University of Ulm), Ulm
- Italy (7):
  - University Polyclinic Hospital "G. Martino", Messina
  - Humanitas Research Hospital IRCCS Istituto Clinico Humanitas, Milan
  - Hospital San Raffaele, Milan
  - Azienda Ospedaliero Universitaria di Modena - Struttura Complessa di Gastroenterologia, Modena
  - Sacred Heart Don Calabria, Negrar
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - University Polyclinic Foundation "Agostino Gemelli", Rome
- Poland (11):
  - Specialist Gastrology Centre GASTROMED, Bialystok
  - Vita Longa Sp. z.o.o., Katowice
  - MEDRISE Sp. z o.o., Lublin
  - SOLUMED Medical Center, Poznan
  - Endoskopia Sp. z o.o., Sopot
  - H-T. Medical Center, Tychy
  - WIP Warsaw IBD Point, Warsaw
  - WSD Medi Clinical Sp. z o.o., Warsaw
  - Planetmed Sp. z o.o., Wroclaw
  - VISTAMED, Wroclaw
  - ETG Zamość, Zamość
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No